CLINICAL TRIAL: NCT05342532
Title: High-Dose Dual Therapy vs Standard Triple Therapy for Treatment-Naïve H. Pylori: A Prospective Randomized Control Trial in a Diverse Urban New York City Population
Brief Title: High Dose Dual Therapy vs Clarithromycin Triple Therapy for Treatment Naive H Pylori Infection in an Urban Population
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Ilan S Weisberg, Assistant Professor of Medicine, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-19-01590
Record Dates: First submitted 2022-04-19; First posted 2022-04-22 (Actual); Results first posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01-05

CONDITIONS: Helicobacter Pylori Infection
Keywords: high-dose dual therapy; standard triple therapy; helicobacter pylori eradication; clarithromycin resistance
MeSH Terms: interventions — Amoxicillin; Omeprazole; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- High Dose Dual Therapy (Active Comparator): This regimen includes a 14-day course of amoxicillin 1 g three times daily and omeprazole 40 mg three times daily.
  Interventions: Drug: Amoxicillin; Drug: Omeprazole
- Standard triple therapy (Active Comparator): This regimen includes a 14-day course of clarithromycin 500 mg twice daily, omeprazole 40 mg twice daily, and amoxicillin 1g twice daily.
  Interventions: Drug: Amoxicillin; Drug: Omeprazole; Drug: Clarithromycin

INTERVENTIONS:
Drug: Amoxicillin — 1 g
Drug: Omeprazole — 40 mg. Patients were asked to take omeprazole one hour prior to food intake, while antibiotics were taken after meals.
Drug: Clarithromycin — 500 mg twice daily
  Arms: Standard triple therapy

SUMMARY:
A phase 4 prospective, randomized, open-label clinical trial evaluating the efficacy of high dose dual therapy vs standard triple therapy in a diverse, urban New York City population.

DETAILED DESCRIPTION:
All patients, at least 18 years of age, with a chief complaint of dyspepsia and documented treatment-naïve HP infection diagnosed on UBT, esophagogastroduodenoscopy (EGD) with HP biopsy, or SAT were recruited for the study. Dyspepsia was defined as persistent or recurrent abdominal pain for at least one month. All subjects who met inclusion criteria were randomly assigned by a computerized system to one of two treatment groups: standard triple therapy (STT) or high-dose dual therapy (HDDT). After patient randomization, all potential side effects were discussed. Education regarding the importance of adherence to complete the full 14 day regimen was provided. Patients were provided an electronic prescription for the respective assigned regimen along with a medication log to self-report drug compliance. The patients were asked to record medication compliance and report any adverse events to research personnel.

After completion of their assigned regimen, subjects were scheduled for a post-treatment visit, 4 weeks after completion of the study. During this period, patients were asked to abstain from taking PPI's to avoid false negative eradication testing. At the post-treatment visit, a medication log and empty pill bottles were brought in to ascertain compliance (defined as completing at least 90% of all prescribed medications).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Treatment-naïve
* Clinical diagnosis of helicobacter pylori infection based on urea breath test, endoscopy or stool antigen test
* Subject willing to participate and able to provide informed consent.

Exclusion Criteria:

* Prior helicobacter pylori treatment failure
* Antibiotic exposure within the past 4 weeks of helicobacter pylori diagnosis
* Pregnancy or breastfeeding
* Penicillin allergy
* History of active or non-gastric malignancy
* Severe illness requiring hospitalization during treatment period
* Starting additional antibiotic while on treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Weisberg, MD, MSc, Principal Investigator — Mount Sinai Beth Israel
Locations (1):
- Mount Sinai Union Square Division of Digestive Diseases, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: Anyone who wishes to access the data. Any purpose. Data are available indefinitely at (Link to be included in the URL field below).

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High Dose Dual Therapy | Standard Triple Therapy
Started | 58 | 54
Completed | 43 | 19
Not Completed | 15 | 35
Not completed — Adverse Event | 5 | 20
Not completed — Lost to Follow-up | 10 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose Dual Therapy | Standard Triple Therapy | Total
Number analyzed (Participants) | 58 | 54 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (15) | 52.7 (14.6) | 51 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 27 | 55
  Male | 30 | 27 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 28 | 54
  Not Hispanic or Latino | 32 | 26 | 58
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participant With Eradication of Disease
Description: The number of participants with eradication after high dose dual therapy vs clarithromycin triple therapy after treatment.
Time Frame: end of study at 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Dual Therapy | Standard Triple Therapy
Number analyzed (Participants) | 58 | 54
Participants | 37 | 42

2. Secondary Outcome: Number of Participants With Protocol Specific Adverse Events
Description: Patient tolerability determined by adverse event rates noted by the presence of abdominal pain, diarrhea, dysgeusia, nausea, vomiting, dysphagia
Time Frame: end of study at 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Dual Therapy | Standard Triple Therapy
Number analyzed (Participants) | 58 | 54
Participants | 5 | 20

3. Secondary Outcome: Number of Participants Completing at Least 90% of All Prescribed Medications
Description: Patients were provided a medication log to self-report drug compliance. After completion of their assigned regimen, subjects were scheduled for a post-treatment visit, 4 weeks after completion of the study. At the post-treatment visit, a medication log and empty pill bottles were brought in to ascertain compliance (defined as completing at least 90% of all prescribed medications).
Time Frame: end of study at 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose Dual Therapy | Standard Triple Therapy
Number analyzed (Participants) | 58 | 54
Participants | 58 | 54

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | High Dose Dual Therapy | Standard Triple Therapy
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/54
Other Adverse Events (participants affected / at risk) | 5/58 | 20/54
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose Dual Therapy (N=58) | Standard Triple Therapy (N=54)
Abdominal pain (Gastrointestinal disorders) | 3 | 7
Diarrhea (Gastrointestinal disorders) | 1 | 2
Dysguesia (Gastrointestinal disorders) | 0 | 4
Nausea (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 5
Dysphagia (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-01-02): https://cdn.clinicaltrials.gov/large-docs/32/NCT05342532/Prot_000.pdf